CLINICAL TRIAL: NCT06750289
Title: BRISOTE: A Multicentre, Randomised, Double-Blind, Parallel Group, Active-Controlled, Phase 3b Study to Evaluate the Efficacy and Safety of Benralizumab 30 mg SC in Eosinophilic Asthma Patients Uncontrolled on Medium-Dose Inhaled Corticosteroid Plus Long-acting β2-Agonist.
Brief Title: Randomised Clinical Trial to Investigate Efficacy and Safety of Benralizumab 30 mg SC as an add-on Therapy in Uncontrolled Eosinophilic Asthma Patients Treated With Medium-dose ICS-LABA Compared to Conventional Escalation to High-dose ICS-LABA Treatment
Acronym: BRISOTE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3250C00101
Record Dates: First submitted 2024-11-20; First posted 2024-12-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Eosinophilic Asthma
Keywords: Eosinophilic Asthma;; Benralizumab,; FASENRA,; Medium-Dose Inhaled Corticosteroid,; Long-acting β2-Agonist
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomised 1:1 to one of the following arms:
  * Medium-dose ICS-LABA + benralizumab
  * High-dose ICS-LABA + placebo (benralizumab)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Benralizumab and placebo will be supplied in identical Accessorised pre-filled syringe (APFS). Medium and high dose ICS-LABA will be supplied in identical inhalers, as appropriate for US and ex-US markets, and the maximum daily dose is the same for the 2 Investigational products (IPs) (2 doses/day).
  Participants are not aware of the dose levels to which they are assigned. The Interactive Response Technology / Randomisation and Trial Supply Management (IRT/RTSM) will provide to the investigator(s) or pharmacist(s) the kit identification number to be allocated to the participant at the dispensing visit.
  Routines for this will be described in the IRT/RTSM user manual that will be provided to each centre.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Medium-dose ICS-LABA + benralizumab (Active Comparator): Participants will be randomised 1:1 to one of the 2 study arms. Participants will receive up to 7 SC injections during study, with the first 3 doses administered every 4 weeks and then subsequent doses every 8 weeks.
  Interventions: Combination Product: ICS-LABA; Combination Product: benralizumab
- High-dose ICS-LABA + placebo (Active Comparator): Participants will be randomised 1:1 to one of the 2 study arms. Participants will receive up to 7 SC injections during study, with the first 3 doses administered every 4 weeks and then subsequent doses every 8 weeks.
  Interventions: Combination Product: ICS-LABA; Combination Product: Placebo for Benralizumab

INTERVENTIONS:
Combination Product: ICS-LABA — ICS-LABA inhalation
Combination Product: benralizumab — Benralizumab. SC injection.
  Arms: Medium-dose ICS-LABA + benralizumab
Combination Product: Placebo for Benralizumab — Placebo for Benralizumab (aka, "placebo"). SC injection.
  Arms: High-dose ICS-LABA + placebo

SUMMARY:
This study evaluates the efficacy and safety of benralizumab as an add-on therapy in uncontrolled eosinophilic asthma participants treated with medium-dose ICS-LABA compared to the conventional treatment step of escalation of inhaled therapy to high-dose ICS-LABA.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-controlled, parallel group global study designed to investigate the efficacy and safety of adding fixed-dose benralizumab (30 mg), administered subcutaneously (SC) every 4 weeks for the first 3 doses and then every 8 weeks for participants with a history of eosinophilic asthma, who remain uncontrolled on medium-dose Inhaled corticosteroid-Long-acting β2-agonists (ICS-LABA) with or without other asthma controller(s) (with the exception of oral corticosteroids), compared to the conventional treatment step of escalation of inhaled therapy to high-dose ICS-LABA plus placebo (benralizumab).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Participant must be 12 to 75 years of age
* Documented history of physician-diagnosed asthma requiring treatment with at least medium-dose ICS (> 250 μg fluticasone dry powder formulation equivalents total daily dose) and a LABA, for at least 12 months prior to Visit (V) 1.
* Documented treatment with medium-dose ICS and LABA for at least 3 months prior to Visit 1 with or without additional asthma controllers (excluding oral corticosteroids).
* Weight of ≥ 35 kg.
* Pre-Bronchodilator (BD) Forced expiratory volume in 1 second (FEV1) of ≤ 90% predicted
* Documented at least 2 asthma exacerbations in the 12 months prior to the date of informed consent.
* ACQ-6 score ≥ 1.5 at Visit 1, plus at least once in the run-in period (from V2 to V3) and at V3.
* Evidence of asthma as documented by excessive variability in lung function, as defined in the protocol.
* Peripheral blood eosinophil count of ≥ 150 cells/μL, as defined in the protocol.
* At least 70% compliance with usual asthma controller ICS-LABA during run-in period (from Visit 2 to Visit 3) based on asthma daily diary.

Exclusion Criteria:

* Important pulmonary disease other than asthma at the discretion of the investigator, or ever been diagnosed with pulmonary or systemic disease, other than asthma, which are associated with elevated peripheral eosinophil counts.
* Asthma exacerbation requiring use of Systemic corticosteroids (SCS), or acute upper/lower respiratory infection that requires antibiotics or antiviral medication within 30 days prior to the date informed consent is obtained or during the screening/run-in period
* Any unstable disorder that in the opinion of the investigator could affect the study according to the study protocol.
* Clinically significant chronic or ongoing active infections requiring systemic treatment (at investigator's discretion)
* Concurrent participation in another clinical study with an IP or a post-authorisation safety study.
* History of alcohol or drug abuse within 12 months prior to the date informed consent is obtained.
* Current smokers or former smokers with a smoking history ≥ 10 pack-years. Former smokers must have stopped for at least 6 months prior to Visit 1 to be eligible.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-11-02 (Estimated); Study Completion 2027-11-02 (Estimated)

PRIMARY OUTCOMES:
Annualized asthma exacerbation rate | Baseline through Week 48
  To assess asthma exacerbation rate.

SECONDARY OUTCOMES:
Change in Saint George's Respiratory Questionnaire (SGRQ) total score | Baseline through Week 48
  The SGRQ is a 50-item ePRO instrument developed to measure the health status of participants with airway obstruction disease. The questionnaire is divided into 2 parts: Part 1 consists of 8 items that pertain to the severity of respiratory symptoms in the preceding 4 weeks, and Part 2 consists of 42 items related to the daily activity and psychosocial impacts of the individual's respiratory condition. The SGRQ yields a total score and 3 component scores (symptoms, activity, and impacts). The total score indicates the impact of disease on overall health status. This total score ranges from 0 to 100 with 0 indicating the best possible health status and 100 representing the worst possible health status
Change in pre-bronchodilator FEV1 | Baseline through Week 48
  Lung function is assessed by FEV1 which was measured by spirometry. Spirometry will be performed by the Investigator or authorized delegate according to American Thoracic Society /European Respiratory Society guidelines.
Change in Asthma control questionnaire (ACQ) scale score. | Baseline through Week 48.
  The ACQ-6 is a shortened version of the full 7-item ACQ questionnaire, which assesses asthma symptoms (nighttime awakening, symptoms on awakening, activity limitation, shortness of breath, wheezing, SABA use) but omits the FEV1 measurement from the original ACQ-7 assessment. Participants are asked to recall how their asthma has been during the previous week by responding to 6 symptom questions. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The total ACQ-6 score is the mean of the responses.
  The effect of benralizumab will be evaluated with the change from baseline in ACQ-6 to End of treatment (week 48) and over the treatment period.
Time to first asthma exacerbation | Baseline through Week 48.
  Time to the first occurrence of asthma exacerbation post randomisation.
Annualized asthma exacerbation rate associated with an emergency/urgent care visit or a hospitalization | Baseline through Week 48.
  The annualized exacerbation rate is based on unadjudicated exacerbation reported by the investigator that are associated with an emergency room/urgent care visit or a hospitalization adjusted by the time of follow-up.
Number and proportion of participants that meet each component of a 4-component clinical remission composite | Week 24 and Week 48.
  * Number and proportion of participants that meet each component of a 4-component clinical remission composite (no exacerbations; no mOCS use; ACQ-6 < 1.5); and stable FEV1 (defined as change from baseline in FEV1 > -100 mL) at Week 24 and EOT.
  * Number and proportion of participants that meet 0, 1, 2, 3 and all 4 components of the composite remission endpoint at Week 24 and EOT.
Safety Adverse Event (AEs), Serious Adverse Event (SAEs), Adverse event leading to treatment discontinuation (DAEs.) | Baseline through Week 48.

CONTACTS AND LOCATIONS:
Locations (126):
- United States (26):
  - Research Site, Chandler, Arizona
  - Research Site, Sun City, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Inglewood, California
  - Research Site, Newport Beach, California
  - Research Site, Pasadena, California
  - Research Site, Denver, Colorado
  - Research Site, Cape Coral, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Ann Arbor, Michigan
  - Research Site, Henderson, Nevada
  - Research Site, Northfield, New Jersey
  - Research Site, New Hyde Park, New York
  - Research Site, The Bronx, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, DuBois, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Greenville, South Carolina
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
- Bulgaria (4):
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Canada (8):
  - Research Site, Edmonton, Alberta
  - Research Site, Kamloops, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Sainte-Foy, Quebec
- China (16):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Huizhou
  - Research Site, Jinan
  - Research Site, Qinhuangdao
  - Research Site, Shanghai
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xuzhou
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
- France (9):
  - Research Site, Bayonne
  - Research Site, Créteil
  - Research Site, La Tronche
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Pessac
  - Research Site, Suresnes
  - Research Site, Toulouse
  - Research Site, Villeurbanne
- Germany (13):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Cottbus
  - Research Site, Delitzsch
  - Research Site, Geesthacht
  - Research Site, Landsberg
  - Research Site, Lübeck
  - Research Site, Mönchengladbach
  - Research Site, München
  - Research Site, München-Pasing
  - Research Site, Neu-Isenburg
  - Research Site, Wiesbaden
  - Research Site, Witten
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, Pok Fu Lam
  - Research Site, Shatin
- Ireland (4):
  - Research Site, Ballinasloe
  - Research Site, Cork
  - Research Site, Dublin
  - Research Site, Moneymore
- Italy (13):
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Brescia
  - Research Site, Cagliari
  - Research Site, Catanzaro
  - Research Site, Genoa
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Montebelluna
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Verona
- Research Site, Lørenskog, Norway
- Spain (16):
  - Research Site, Alcorcón
  - Research Site, Alzira (Valencia)
  - Research Site, Badalona
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Cáceres
  - Research Site, Granada
  - Research Site, Jerez de la Frontera
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Marbella
  - Research Site, Málaga
  - Research Site, Mérida
  - Research Site, Palma de Mallorca
  - Research Site, Santander
- Switzerland (5):
  - Research Site, Aarau
  - Research Site, Basel
  - Research Site, Lausanne
  - Research Site, Sankt Gallen
  - Research Site, Sion
- United Kingdom (8):
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Bristol
  - Research Site, Chorley
  - Research Site, Leeds
  - Research Site, Nottingham
  - Research Site, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/